CLINICAL TRIAL: NCT02409836
Title: A Study to Assess the Ingestion of Dentifrice by Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 000393
Record Dates: First submitted 2015-03-24; First posted 2015-04-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Healthy Individuals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Crest Cavity Protection (Active Comparator): Marketed Dentifrice
  Interventions: Drug: Marketed Dentifrice
- Crest for Kids Hawaiian Punch Paste (Active Comparator): Marketed Dentifrice
  Interventions: Drug: Marketed Flavored Dentifrice
- Crest for Kids Bubble Gum Paste (Active Comparator): Marketed Dentifrice
  Interventions: Drug: Marketed Flavored Dentifrice

INTERVENTIONS:
Drug: Marketed Dentifrice — Marketed Dentifrice
  Arms: Crest Cavity Protection
Drug: Marketed Flavored Dentifrice — Hawaiian Punch Flavored
  Arms: Crest for Kids Hawaiian Punch Paste
Drug: Marketed Flavored Dentifrice — Bubble Gum Flavored
  Arms: Crest for Kids Bubble Gum Paste

SUMMARY:
The objective of this study was to examine the amount of dentifrice ingested and used by various age groups of children.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 2 and 12, inclusive
* Be healthy, with no illness that, in the judgment of the investigator or examining dentist, would interfere with the conduct of the test
* Be currently, and have been for at least three months immediately prior to the start of the study, brushing (or being brushed by care giver) their teeth on a daily basis
* Have parent/guardian complete and return the consent form

Exclusion Criteria:

* Have diabetes
* Be on dialysis
* Have an oral health condition that, in judgment of investigator or study medical personnel, could interfere with the conduct of the study.
* Wear metal braces
* Have an incomplete or missing consent form

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 1993-05; Primary Completion 1993-07 (Actual); Study Completion 1993-07 (Actual)

PRIMARY OUTCOMES:
Level of dentifrice ingested and used by various age groups of children. | 10 weeks

SECONDARY OUTCOMES:
Dentifrice ingestion amount as a function of dentifrice flavor and age of participants. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John E Wild, Principal Investigator — HIlltop Research Inc.
Locations (1):
- Hill Top Research, Inc., Cincinnati, Ohio, United States